CLINICAL TRIAL: NCT07054892
Title: EntoQuaVie - Assessment of the Quality of Life of Patients Visiting the Emergency Department of the Saint-Brieuc Hospital Following an Ankle Sprain: A Follow-up-based Evaluation Considering the Severity Grade of the Ankle Sprain
Brief Title: Assessment of the Quality of Life of Patients Visiting the Emergency Department of the Saint-Brieuc Hospital Following an Ankle Sprain
Acronym: EntoQuaVie
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_CHSB_EntoQuaVie; 2024-A02526-41 (Other: ID RCB)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ankle Injuries; Treatment Outcome
Keywords: ankle injuries; emergency department; patient follow-up
MeSH Terms: conditions — Ankle Injuries; Emergencies | interventions — Activities of Daily Living

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with ankle sprain: Participants presenting to the emergency department of Saint-Brieuc for an ankle sprain
  Interventions: Behavioral: FAAM - Activities of Daily Living (ADL) Subscale

INTERVENTIONS:
Behavioral: FAAM - Activities of Daily Living (ADL) Subscale — The FAAM score is scientifically validated and allows for the assessment of foot and ankle functional ability

SUMMARY:
Lateral ankle sprains account for nearly 6,500 emergency department visits per day in France. They are clinically classified into three grades, which can be assessed approximately 3-5 days after an acute sprain. However, this classification remains somewhat approximate, with only mild and severe sprains being reliably identified.

When it comes to immobilization, if weight-bearing is possible, treatment options include an elastic ankle brace for mild sprains, taping, or a semi-rigid orthosis known as a "stabilizing" brace. It is worth noting that, according to Rodineau and Besch, the preferred form of immobilization is the semi-rigid orthosis. In cases of severe sprains where weight-bearing is not possible, rigid immobilization may be used.

To date, few thesis-level studies have focused on trauma care and the outpatient follow-up of ankle sprains. Two studies from the early 2010s assessed general practice management of trauma using questionnaires-one in Seine-Maritime and another in Bouches-du-Rhône. The latter study found that 96.7% of surveyed physicians reported managing all types of sprains. In the Seine-Maritime study, half of the physicians systematically followed up on ankle sprains, while the other half only did so if the patient's condition worsened. It was also found that nearly 47% of physicians referred their patients directly to emergency departments. This pathway was more frequently chosen by urban practitioners or those without specific training in trauma care.

Except in certain predefined cases depending on the hospital, there is currently no systematic follow-up for ankle sprains in emergency departments. Most patients are redirected toward follow-up in outpatient care.

The objective of this research project is to assess the recovery of baseline quality of life in participants who consulted the emergency department of Saint-Brieuc for an ankle sprain, three months after the injury. The evaluation will take into account the type of follow-up care (physician, physiotherapist) as well as the severity of the sprain.

DETAILED DESCRIPTION:
The FAAM-ADL questionnaire is a self-assessment tool and will be completed for the first time upon the participant's arrival at the emergency department. The responses will be based on the participant's recollection of their functional ability and quality of life prior to the ankle injury.

A second self-assessment will be conducted at the 3-month mark, using the same FAAM-ADL scale, either by email or phone. This time, the questionnaire will focus on their current functional ability and quality of life. By comparing these two sets of responses, it will be possible to evaluate the degree of recovery three months after the ankle sprain, relative to their pre-injury baseline.

The severity grade of the sprain will be determined based on the clinical data recorded by the physician during the initial emergency consultation, following review of the medical records by the coordinating investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ankle trauma
* Initial consultation at the emergency department of Saint-Brieuc

Exclusion Criteria:

* Surgical treatment following the trauma
* Fracture resulting from the trauma
* Ligament or bone injury to either lower limb (knee, hip, ankle) occurring within 6 months prior to the trauma
* Injury to another joint during the trauma with functional impairment
* Adult under legal protection (guardianship, trusteeship, or judicial protection) or deprived of liberty
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants presenting to the emergency department of Saint-Brieuc for an ankle sprain.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
FAAM ADL questionnaire | At inclusion in the study and 3 months later
  The FAAM-ADL questionnaire is the first subscale of the FAAM questionnaire. It consists of 21 items and is used to assess activities of daily living. Each item is rated on a scale from 0 to 4 (0: unable to perform the activity; 4: no difficulty performing the activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Brieuc - Paimpol - Tréguier, Saint-Brieuc, France

IPD SHARING:
Plan to Share IPD: Undecided